CLINICAL TRIAL: NCT06670820
Title: The Effects of Intermittent Theta-burst Stimulation on Cognitive Function in Patients with Mild Cognitive Impairment and Mild Alzheimer's Disease and the Role of Brain-Derived Neurotrophic Factor
Brief Title: ITBS in MCI and Mild AD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Yu-Kai Lin, Tri-Service General Hospital, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: A202305164
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment (MCI); Mild Alzheimer Disease
Keywords: rTMS; iTBS; Mild Cognitive Impairment; Mild Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active iTBS for Patients With MCI or AD (Active Comparator): The patient will receive one daily rTMS session for 10 days of iTBS, delivered through an H-coil applied to the left dorsolateral prefrontal cortex. The TBS frequency parameters consist of 3-pulse 50-Hz bursts every 200 ms at 5 Hz, and the intensity will be set at 80% of the active motor threshold (AMT). A single session of iTBS contains 2 s of TBS repeated every 10 s for 20 times.
  Interventions: Device: Active rTMS
- Sham iTBS for Patients With MCI or AD (Sham Comparator): Sham stimulation will be delivered 10 sessions.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — iTBS targeting the left dorsolateral prefrontal cortex (DLPFC) per session, total10 sessions
  Arms: Active iTBS for Patients With MCI or AD
Device: Sham rTMS — sham iTBS targeting the left dorsolateral prefrontal cortex (DLPFC) per session, total 10 sessions
  Arms: Sham iTBS for Patients With MCI or AD

SUMMARY:
This study aims to examine the effects of iTBS on cognitive function in individuals with MCI or mild AD, with a secondary objective of exploring prefrontal TBS mechanisms for cognitive function and the effect of iTBS on BDNF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MCI (overall Clinical Dementia Rating of 0.5)
* Clinical diagnosis of mild Alzheimer's Disease (overall Clinical Dementia Rating of 0.5 or 1)

Exclusion Criteria:

* History of stroke
* History of uncontrol seizure
* History of significant head trauma followed by persistent neurologic deficit or known structural brain abnormality
* Mental illness
* Drug abuse

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in neurocognitive function test scores (Mini-Mental State Examination；MMSE) between T1 (Day 1) and T2 (Day 14), and the differences between the experimental and control groups. | MMSE will be controlled at baseline before active or sham rTMS, 2 weeks after active and sham rTMS, 3 months after the last treatment
  The mini-mental state examination (MMSE) test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.The MMSE is a standardized cognitive screening test with a possible score of 0-30. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.

SECONDARY OUTCOMES:
Changes in neurocognitive function test scores (Mini-Mental State Examination；MMSE) between T1(Day 1) and T3 (98 ± 14), and the differences between the experimental and control groups. | MMSE will be controlled at baseline (T1: Day 1) before active or sham rTMS, 2 weeks after active and sham rTMS (T2: Day 17 ± 5), 3 months after the last treatment (T3: Day 98 ± 14).
  The mini-mental state examination (MMSE) test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.The MMSE is a standardized cognitive screening test with a possible score of 0-30. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Changes in blood BDNF concentration levels before and after active rTMS and after sham rTMS, as well as the differences between the experimental group and the control group | BDNF will be controlled at baseline ( Day 1) before active or sham rTMS, 2 weeks after active and sham rTMS (Day 17 ± 5).
Side effects between the two groups. | Side effects will be monitored during 2 groups (active and sham) through study completion, an average of 3-4 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Other, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24833712/